CLINICAL TRIAL: NCT02713269
Title: A Phase II Clinical Trial Evaluating the Efficacy of Combining Thermal Ablation and Spine Stereotactic Radiosurgery for Patients With Spine Metastases With Moderate to Severe Epidural Involvement
Brief Title: Thermal Ablation and Spine Stereotactic Radiosurgery in Treating Patients With Spine Metastases at Risk for Compressing the Spinal Cord
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0223; NCI-2016-00683 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0223 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Malignant Digestive System Neoplasm; Metastatic Head and Neck Carcinoma; Metastatic Kidney Carcinoma; Metastatic Malignant Neoplasm in the Spine; Metastatic Malignant Neoplasm of Unknown Primary; Metastatic Melanoma; Prostate Carcinoma Metastatic in the Bone; Sarcoma; Solid Neoplasm; Spinal Cord Compression; Stage IV Breast Cancer AJCC v6 and v7; Stage IV Lung Non-Small Cell Cancer AJCC v7; Thyroid Gland Carcinoma
MeSH Terms: conditions — Gastrointestinal Neoplasms; Carcinoma, Renal Cell; Neoplasms, Unknown Primary; Melanoma; Sarcoma; Spinal Cord Compression; Thyroid Neoplasms | interventions — Radiosurgery; Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No

ARMS (1):
- Treatment (thermal ablation, SSRS) (Experimental): Patients undergo thermal ablation and CT-guided SSRS via intensity-modulated radiation therapy on different dates within a 1-14 day window. The order of treatment is at the doctor's discretion.
  Interventions: Procedure: Computed Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Radiosurgery; Procedure: Thermal Ablation Therapy

INTERVENTIONS:
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; computerized tomography; CT; CT SCAN; tomography
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Radiosurgery — Undergo CT-guided SSRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; stereotactic radiation therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
Procedure: Thermal Ablation Therapy — Undergo thermal ablation therapy
  Other Names: thermal ablation

SUMMARY:
This phase II clinical trial studies how well thermal ablation and spine stereotactic radiosurgery work in treating patients with cancer that has spread to the spine (spine metastases) and is at risk for compressing the spinal cord. Thermal ablation uses a laser to heat tumor tissue and helps to shrink the tumor by destroying tumor cells. Stereotactic radiosurgery delivers a large dose of radiation in a short time precisely to the tumor, sparing healthy surrounding tissue. Combining thermal ablation with stereotactic radiosurgery may be a better way to control cancer that has spread to the spine and is at risk for compressing the spinal cord.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To document the rate of local control at 6 months in patients who receive a combination of thermal ablation and stereotactic spine radiosurgery (SSRS) for spine metastases with moderate to severe epidural involvement.

SECONDARY OBJECTIVES:

I. To determine local control at 1, 3, 9, 12, 18, and 24 months, and to compare to a historical control where patients received only SSRS at these time points and at 12 months.

II. To document the extent of epidural tumor regression at 1, 3, 6, 9, 12, 18 and 24 months.

IIa. Calculate decrease in epidural tumor volume (by volumetric measurements). IIb. Calculate increase in thecal sac patency (by volumetric measurements and according to Bilsky method).

III. To determine overall survival at 6, 12, 18, and 24 months. IV. To assess changes in muscle strength, location and severity of spinal-related pain, sensory function, ability to ambulate, and neurological grading at 1, 3, 6, 9, 12, 18, and 24 months compared with pretreatment baselines.

V. To assess the effect of treatment on quality of life (QOL), measured at 1 month and every 3 months after with validated outcome measure tools.

VI. To describe adverse side effects after treatment and to descriptively correlate those effects with radiographic findings, pain control, and quality of life.

OUTLINE:

Patients undergo thermal ablation and computed tomography (CT)-guided SSRS via intensity-modulated radiation therapy on different dates within a 1-14 day window. The order of treatment is at the doctor's discretion.

After completion of study treatment, patients are followed up at 1, 3, 6, 9, and 12 months and then every 6 months.

ELIGIBILITY:
Inclusion:

* At least 18 years of age.
* Histologic diagnosis of solid malignant tumor (not one of the more radiosensitive histologic subtypes, see Exclusion Criteria), including but not limited to non-small cell lung cancer, breast, prostate, renal cell, melanoma, gastrointestinal, sarcoma, thyroid, head and neck primary, and unknown primary tumors.
* Quantification of the degree of epidural spinal cord compression as grade 1C, 2, or 3 by MRI, with and without contrast sequences. Axial T2 sequence is encouraged but not required.
* The vertebral body site to be treated must be located from T2-T12.
* No more than 3 contiguous or discontiguous vertebral levels involved with metastasis in the spine to be irradiated in a single session or 3 sessions.
* Motor strength >/=4 out of 5 in extremity or extremities affected by the level of the spinal cord compression (see section 4 for grading method).
* ECOG performance status </=2 or Karnofsky performance status (KPS) >/=50
* Life expectancy >3 months.
* Inoperable disease because of patient refusal, neurosurgical evaluation, or any other medical reasons.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) before study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Prior conventional radiation to the same site is allowed as long as there is a greater than 3 months interval.
* All patients must sign informed consent forms verifying that they are aware of the investigational nature of this study in keeping with the rules and policies of MD Anderson Cancer Center. The only acceptable consent form is one approved by the MD Anderson institutional review board.
* Patients who do not have other options of treatment, based on consensus recommendation of the multidisciplinary spine SRS (SSRS) tumor board. Patients will have an appropriate medical oncologist for their disease.

Exclusion:

* Primary tumors of radiosensitive histology (lymphoma, multiple myeloma, small cell carcinoma, germ cell tumors), as conventional radiation is likely to be effective in such cases.
* Prior conventional irradiation of the spine site and level to be treated with an interval shorter than 3 months.
* Lesions located outside of the spinal segments of T2 to T12.
* Prior surgery to the same levels of spine.
* Inability to lie flat on a treatment table for >60 minutes.
* Unable to undergo MRI of the spine
* Pregnancy (because radiation has the potential for teratogenic or abortifacient effects).
* Frank cord compression or cord compression from bone components or configuration and acute neurological deficits (defined as motor strength <4/5 in extremity or extremities affected by the level of the spinal cord compression).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2027-10-28 (Estimated); Study Completion 2027-10-28 (Estimated)

PRIMARY OUTCOMES:
Local tumor control rate | At 6 months
  Kaplan-Meier estimates will be used.

SECONDARY OUTCOMES:
Local tumor control | Up to 24 months
  Kaplan-Meier estimates will be used. Time to local failure will be monitored continuously using a Bayesian method. Cumulative incidence of local failure will be estimated failure treating death without failure as a competing risk. Propensity score analyses will be used to compare the thermal ablation cohort with a historical cohort where patients received only stereotactic spine radiosurgery (SSRS).
Epidural control assessed by volumetric measurements | Up to 24 months
  Extent of epidural tumor regression be determined by change in epidermal tumor volume and change in thecal sac patency (by volumetric measurements and according to Bilsky method). Kaplan-Meier estimates will be used. Cumulative incidence of epidural failure will be estimated failure treating death without failure as a competing risk. Propensity score analyses will be used to compare the thermal ablation cohort with a historical cohort.
Overall survival | Up to 24 months
  Kaplan-Meier estimates will be used.
Changes in symptoms assessed by physical examination | Baseline to 24 months
  The Physical exam includes general exam, (HEENT) Head, Eye, Ear, Nose and Throat evaluation, chest, heart, abdomen and extremities exam. Combined with the neurotically examination results, changes at 1, 3, 6, 9, 12, 18, and 24 months will be compared with pretreatment baselines. Patients with negative changes will be evaluated by the neurosurgeon and radiation oncologist to determine if the change is related to a local failure/complication or to progression of systemic disease. Kaplan-Meier estimates will be used.
Changes in symptoms assessed by neurological examination | Baseline to 24 months
  The neurological exam includes (1) mental status (tested through history taking), (2) cranial nerves (Observation of eyes, face, voice, and coordination during history taking and as patient moves about the exam room. Look for extraneous movements), (3) motor system (visual inspection, tone, muscle strength and endurance, assigned score of 0-5 for each muscle, a score of 0 would mean no muscular contraction, and a score of 5 would mean movement against full resistance, normal strength), (4) reflexes, (5) sensory system (vibration in toes; pinprick in feet; (6) coordination (Truncal stability, fine finger movement, toe tapping, finger-nose-finger, heel-knee-shin), and (7) station and gait (Gait including arising from chair without hands, walking on toes, heels, and heel to toe). Kaplan-Meier estimates will be used.
Changes in quality of life (QOL) assessed by the MD Anderson Symptom Inventory Spine Tumor form | Baseline to 24 months
  Participants are asked to recall symptom severity and interference during the past 24 hours. Part I, The severity of the symptoms, including pain, fatigue, nausea, disturbed sleep, short of breath etc. Part II, How have the symptoms interfered with patient life, including mood, work, relations with other people etc. Part I, range 0-10. A score of 0 would mean the symptom is not present and a score of 10 means the symptom is as bad as you can imagine). Part II, range 0-10 (A score of 0 would mean the symptom did not interfere; A score of 10 means the symptom has interfered completely).
Changes in quality of life (QOL) assessed by Brief pain inventory (BPI) form | Baseline to 24 months
  Participants are asked to assess the severity of pain and the impact of pain on daily functions. Severity of pain, including the pain location, worst pain in last 24 hours, least pain in last 24 hours, pain on average and pain right now. Range 0-10. A score of 0 would mean no pain and a score of 10 means the pain is as bad as you can imagine. Pain medications, amount of pain relief in the past 24 hours, and impact of pain on daily function, including general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life, and Range 0-10.
Changes in quality of life (QOL) assessed by SF-12 healthy survey (v2) | Baseline to 24 months
  Participants are asked to twelve questions that measure eight health domains to assess physical and mental health. Physical health-related domains include General Health (GH), Physical Functioning (PF), Role Physical (RP), and Body Pain (BP). Mental health-related scales include Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH). 3 and 5 point Likert scale is used in the survey. Two summary scores of the SF-12v2-physical and mental health-using the weighted means of the eight domains. Descriptive statistics will be used to summarize pain relief and quality of life at each follow-up visit, which will be the changes in scores from baseline to each assessment visit. Time to maximum pain relief will be the time from the day of thermal ablation until the lowest pain score for average pain after radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org